CLINICAL TRIAL: NCT05355389
Title: Cognitive-motor Telerehabilitation in Multiple Sclerosis
Brief Title: Cognitive-motor Telerehabilitation in MS
Acronym: CoMoTeMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: National MS Center Melsbroek (Other); Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CoMoTeMS; 1SD5322N (Other Grant/Funding Number: Fonds Wetenschappelijk Onderzoek (FWO))
Record Dates: First submitted 2022-04-14; First posted 2022-05-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; cognitive rehabilitation; cognitive-motor rehabilitation; telerehabilitation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either the cognitive-motor, the cognitive or the motor telerehabilitation group, stratified by baseline activity level and cognition.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded: patients will not be made aware of the rationale and predictions of the study. The teleconsultations will be carried out by a trained MS nurse, while the baseline and follow-up testing and analyses are carried out by an investigator who is blinded to the treatment allocation of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive-motor training group (Experimental)
  Interventions: Behavioral: Cognitive training; Behavioral: Motor training
- Cognitive training group (Active Comparator)
  Interventions: Behavioral: Cognitive training
- Motor training group (Active Comparator)
  Interventions: Behavioral: Motor training

INTERVENTIONS:
Behavioral: Cognitive training — For the cognitive treatment intervention the widely used cognitive training program RehaCom will be used. This is a computer-aided program with more than 30 modules focusing on different domains of cognition. RehaCom has shown improvements in verbal learning, visuospatial memory, information processing speed, attention, executive functions, depression, fatigue and quality of life in PwMS (PMID 31927200, 28116167, 19825502, 23192417). Patients will train on their home computer without direct therapist supervision, using three RehaCom modules that are focused on improving working memory. Both patients in the combined intervention and the cognitive intervention group will be doing a 45-minute computer session respectively one and two days per week for a total of 12 weeks.
  Other Names: BrainStim
  Arms: Cognitive training group; Cognitive-motor training group
Behavioral: Motor training — For the motor treatment intervention a patient-tailored aerobic training program will be used. Based on their baseline physical activity level patients can choose out of a number of aerobic activities of either mild, moderate or strenuous intensity, with a total training time of 90 minutes for the motor intervention group and 45 minutes for the combined intervention group, divided over at least two training sessions per week of at least 15 minutes per session. The training will be carried out individually at home, without therapist supervision. All physical activities will be logged using the sport watch equipped with a heart rate sensor and an accelerometer. Training intensity will be assessed using the patient's heart rate and the Rating of Perceived Exertion scale.
  Arms: Cognitive-motor training group; Motor training group

SUMMARY:
The primary goal of this project is providing evidence that a home-based combined cognitive-motor training program improves cognition in persons with multiple sclerosis (MS), compared to single cognitive and motor rehabilitation. Secondary goals are to assess the effects on walking performance and to identify the mechanisms of improvement and predictors of treatment response. The main backbone of this project will be a randomized controlled two-centre clinical trial, in which an at-home computerised cognitive-motor rehabilitation program using telemedicine aimed at improving working memory in persons with MS will be evaluated. Based on the information gathered during this trial, possible mechanisms of improvement will be identified by analysing anatomical and neurophysiological changes on structural MRI and resting-state and task-related EEG before and after rehabilitation. Furthermore, factors that can predict treatment response to the rehabilitation program will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite multiple sclerosis (revised McDonald criteria 2017)
* Expanded Disability Status Scale (EDSS) below 6.0
* Digit span backwards z-score between [-3 and -0.5] standard deviations below the median of the normative values
* Age between 18 and 65
* Able to safely perform motor rehabilitation in the home situation (assessed by rehabilitation physician and/or occupational or physiotherapist)

Exclusion Criteria:

* Cognitive rehabilitation within six months before inclusion
* Inpatient multidisciplinary rehabilitation program within three months before inclusion or planned inpatient program during trial
* Start of or switch in immunomodulator treatment within three months before inclusion
* Less than one month post-exacerbation
* Major psychiatric or medical disorder that could influence cognitive functions
* Combined vision with optimal correction below 0.6 on Snellen Visual Acuity Test
* Unable or unwilling to undergo EEG or MRI
* Refusing informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Digit span backwards | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of working memory

SECONDARY OUTCOMES:
Change in Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of cognition in MS
Change in Corsi backwards | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of working memory
Change in Expanded Disability Status Scale (EDSS) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of disability in MS
Change in 6-Minute Walk Test (6MWT) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of walking performance
Change in 25-Foot Walk Test (25FWT) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of walking performance
Change in 9-Hole Peg Test (9HPT) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of upper extremity function
MRI T1 3D BRAVO scan | 0 weeks, 12 weeks, 24 weeks
  Cortical volume, volumes of white matter and deep grey matter
MRI T2 FLAIR 3D Cube scan | 0 weeks, 12 weeks, 24 weeks
  Lesion volume
Diffusion weighted image (DWI) | 0 weeks, 12 weeks, 24 weeks
  structural connectivity using graph theoretical measures; diffusion tensor image parameters
Synthetic MRI | 0 weeks, 12 weeks, 24 weeks
  Contrast weighted images based on measurements of tissue properties from a single acquisition
resting-state EEG | 0 weeks, 12 weeks
  functional connectivity using graph theoretical measures
task-related EEG - auditory oddball paradigm | 0 weeks, 12 weeks
  functional connectivity using graph theoretical measures, event-related potentials
task-related EEG - adjusted SDMT paradigm | 0 weeks, 12 weeks
  functional connectivity using graph theoretical measures, event-related potentials
task-related EEG - n-back paradigm | 0 weeks, 12 weeks
  functional connectivity using graph theoretical measures, event-related potentials

OTHER OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of anxiety and depression
Change in Fatigue Scale for Motor and Cognitive functions (FSMC) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of fatigue in MS
Change in Visual Analogue Scale (VAS) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  VAS on the impact of perceived cognitive symptoms on daily life
Change in 36-Item Short Form Survey (SF-36) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of quality of life Only Dutch-speaking participants
Change in Multiple Sclerosis Impact Scale-29 (MSIS-29) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of quality of life in MS Only Dutch-speaking participants
Change in Multiple Sclerosis-59 (SEP-59) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of quality of life, combination of SF-36 and MS-specific questions Only French-speaking participants Of note, the French title of this questionnaire is Sclérose En Plaques-59.
Change in Cognitive Leisure Activity Scale (CLAS) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of baseline cognitive activities
Change in Godin Leisure-Time Exercise Questionnaire (GLTEQ) | 0 weeks, 12 weeks, 24 weeks, 64 weeks
  Measure of baseline physical activities

CONTACTS AND LOCATIONS:
Overall Officials: Guy Nagels, Principal Investigator — Vrije Universiteit Brussel, Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - National MS Center Melsbroek, Melsbroek

REFERENCES:
- [Derived] Van Laethem D, Van de Steen F, Kos D, Naeyaert M, Van Schuerbeek P, D'Haeseleer M, D'Hooghe MB, Van Schependom J, Nagels G. Cognitive-motor telerehabilitation in multiple sclerosis (CoMoTeMS): study protocol for a randomised controlled trial. Trials. 2022 Sep 14;23(1):778. doi: 10.1186/s13063-022-06697-9. PMID 36104820